CLINICAL TRIAL: NCT02764710
Title: Randomized Controlled Trial Comparing Long and Short Duration of Antibiotic Prophylaxis for Patients Undergoing Sinus Lift Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Head of Resaerch and Development Department, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TASMC-15-RB-0059-CTIL
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Maxillofacial Surgery
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Short treatment (Experimental): Short course of postoperative treatment: amoxicillin-clavulanate 875mg, one tab twice daily for a total of 2 doses.
  Interventions: Drug: Amoxicillin-Potassium Clavulanate Combination
- Long treatment (Active Comparator): Long course of postoperative treatment: amoxicillin-clavulanate 875mg, one tab twice daily up until and including postoperative day 7.
  Interventions: Drug: Amoxicillin-Potassium Clavulanate Combination

INTERVENTIONS:
Drug: Amoxicillin-Potassium Clavulanate Combination — Short course of postoperative treatment: amoxicillin-clavulanate 875mg, one tab twice daily for a total of 2 doses.
  Long course of postoperative treatment: amoxicillin-clavulanate 875mg, one tab twice daily up until and including postoperative day 7.

SUMMARY:
The optimal use of prophylactic antibiotic therapy to prevent infection after sinus lift and augmentation surgery is unknown. This is a comparative open label interventional trial comparing a standard 7-day course of postoperative treatment with amoxicillin-clavulanate with short antibiotic treatment for up to 24 hours postoperatively. The primary study outcome is the postoperative surgical site infection in the standard versus the short treatment arms. Secondary outcomes are drug-related adverse events and Clostridium difficile infection.

DETAILED DESCRIPTION:
Research rational

The use of antibiotics as prophylaxis for surgical site infection (SSI) is well based in most fields of surgery. The use of prophylactic antibiotics can reduce the rate of post-surgical infections substantially. Nonetheless, overuse of these drugs is likely to expose patients to adverse effects, increase the rate of microbial drug resistance and lead to unnecessary expenses.

In the field of dentistry there are recommendations for prevention of infective endocarditis. The use of antibiotics for SSI in the field of oral and maxillofacial surgery is not well established, with inconsistent and even contradictory recommendations.

Sinus floor lift and augmentation is a common surgical procedure in modern dentistry. It aims to increase the amount of bone in the posterior maxilla, in the area of the premolar and molar teeth, prior to placement of dental implants. The procedure is performed in a per-oral approach; a mucoperiosteal flap is elevated, the lateral boney wall of the sinus is exposed and a window is cut with a surgical bur. The Schneiderian membrane (sinus periost) is separated and lifted from the bone and a bone graft material is placed into the newly created space. The graft material used can be an autograft, an allograft, a xenograft, an alloplast or a combination of these materials.

The rate of post-operative infection after a sinus lift procedure reaches 7%. An evidence based approach for antibiotic prophylaxis for this procedure does not exist. The standard of care is based on clinical experience and protocols for placing dental implants in the jaws bone.

The current protocols include broad spectrum antibiotics aimed at oral bacteria and main pathogens in acute bacterial sinusitis (Streptoccocus pneumoniae, Moraxella catarrhalis, Haemophilus influenzae): amoxicillin+clavulanic acid or clindamycin / clarithromycin+metronidazole for patients with penicillin allergy. According to the common protocol, the antibiotics are given one day prior to surgery or at the day of surgery (one hour before the first cut) and are continued for seven days post-operatively. This practice contradicts the current recommendation for a shortened postoperative course of antimicrobials for less than 24 hours (10). No evidence suggests that prescribing antibiotics beyond 24 hours lowers the rate of SSI. On the other hand, a prolonged prophylactic regimen elevates the risk of Clostridium difficile infection and contributes to antibiotic resistance.

Lindenboom and Van den Akker have demonstrated in 2003 that not administrating prophylactic antibiotics at all prior to bone augmentation elevates the rate of SSI significantly in comparison with a patient who receives antibiotics. On the other hand, our clinical experience shows that short term prophylactic antibiotics (up to 3 days post-operatively) in sinus augmentation surgery and other bone augmentations in the oral cavity do not elevate the risk of SSI. The need to prescribe antibiotics for more than 24 hours post-operatively was never evaluated in a clinical trial.

In the current trial we will test the hypothesis that a short prophylactic regimen does not differ from a prolonged one. On the contrary, we hypothesize that the adverse effects rate will be lower in patients that will receive antibiotics for a short period.

Aim of the study

This is a prospective randomized non-blinded trial which compares a short prophylactic regimen (till on day post-operatively) with a long prophylactic regimen (till seven days post-operatively as acceptable currently) in patients that undergo sinus augmentation surgery.

Study hypothesis: both groups will display similar rates of SSIs.

Materials and methods

The participants will be recruited from patients in Tel-Aviv Medical Center dental clinic that are in need for a unilateral or bilateral sinus augmentation surgery.

The recruited patients will meet the chief investigator for a thorough explanation on the trial, emphasizing the fact that the surgery itself is not the essence of this trial. After signing an informed consent for participating in the trial, the patients will be randomly split into two groups. The recruited patients will receive a prescription for antibiotics and how to take them: amoxicillin-clavulanate 875mg twice a day starting at the morning of surgery. Patient with penicillin allergy will receive a loading dose of clindamycin 300mg, followed by 150mg every 6 hours. The duration of treatment (one day or seven days post-operatively) will be determined according to the group attribution.

The sinus augmentation surgeries will be performed by the attending surgeons at the Oral and Maxillofacial department, according to a unified protocol: a pre-op chlorhexidine 2% rinse, local anesthesia with Lidocaine 2% with adrenalin 1:100000, elevation of a mucoperiosteal flap to expose the lateral wall of the sinus, performing an access window in the bony wall and lifting the sinus membrane, augmentation of the cavity using a xenogeneic and /or allogeneic bone graft substitute and a collagen membrane, placement of dental implants if feasible and suturing of the flap.

Augmenting the cavity with different materials reflects the common practice and based on the fact that these differences do not alter the rate of post-operative complications or dental implants failure in sinus augmentation sites.

Further treatment with dexamethasone, decongestants and pain medications will be administered according to current protocols and are subject to the surgeon's judgment in order to reflect the common practice.

The patients will be evaluated at the following appointed times until the placement/exposure of the dental implants: one week, two weeks, one month, two months, six months. These dates are part of the standard of care as a follow-up after sinus augmentation surgery.

Patients will be withdrawn from the study if they will not attend the follow-up appointments.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient (18 years of age or older) that requires a unilateral or bilateral sinus augmentation surgery.
2. Weight <150 kg.

Exclusion Criteria:

1. Need for prophylactic antibiotics for infective endocarditis.
2. Chronic antibiotics therapy.
3. Special populations: pregnant women, minors and legally incompetent patients.
4. Patients receiving anticoagulants.
5. Non-balanced diabetes mellitus.
6. Immune-suppression: corticosteroids treatment equivalent to 15mg prednisone for at least 14 days in the past month; chemotherapy, TNF inhibitor or drugs that suppress T-cell activity during the past 90 days; HIV infection.
7. Pathology of the maxillary sinus.
8. History of chronic sinusitis.
9. Patients that underwent a Caldwell-Luc procedure.
10. Patients with residual teeth roots at the planned surgical site.
11. A known state of carriage of Methicillin resistant Staphylococcus aureus or Clostridium difficile in the past year.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection rate | 30 days
  Deep or superficial SSI according to CDC/NHSN criteria

SECONDARY OUTCOMES:
Diarrhea | 30 days
  Diarrheal illness reported by patient.
Clostridium difficile infection | 30 days
  Laboratory confirmed C. diff. infection
Adverse event rate | 30 days
  Any reported adverse event

REFERENCES:
- [Background] Young PY, Khadaroo RG. Surgical site infections. Surg Clin North Am. 2014 Dec;94(6):1245-64. doi: 10.1016/j.suc.2014.08.008. Epub 2014 Oct 3. PMID 25440122
- [Background] Wilson W, Taubert KA, Gewitz M, Lockhart PB, Baddour LM, Levison M, Bolger A, Cabell CH, Takahashi M, Baltimore RS, Newburger JW, Strom BL, Tani LY, Gerber M, Bonow RO, Pallasch T, Shulman ST, Rowley AH, Burns JC, Ferrieri P, Gardner T, Goff D, Durack DT; American Heart Association Rheumatic Fever, Endocarditis, and Kawasaki Disease Committee; American Heart Association Council on Cardiovascular Disease in the Young; American Heart Association Council on Clinical Cardiology; American Heart Association Council on Cardiovascular Surgery and Anesthesia; Quality of Care and Outcomes Research Interdisciplinary Working Group. Prevention of infective endocarditis: guidelines from the American Heart Association: a guideline from the American Heart Association Rheumatic Fever, Endocarditis, and Kawasaki Disease Committee, Council on Cardiovascular Disease in the Young, and the Council on Clinical Cardiology, Council on Cardiovascular Surgery and Anesthesia, and the Quality of Care and Outcomes Research Interdisciplinary Working Group. Circulation. 2007 Oct 9;116(15):1736-54. doi: 10.1161/CIRCULATIONAHA.106.183095. Epub 2007 Apr 19. PMID 17446442
- [Background] Anitua E, Aguirre JJ, Gorosabel A, Barrio P, Errazquin JM, Roman P, Pla R, Carrete J, de Petro J, Orive G. A multicentre placebo-controlled randomised clinical trial of antibiotic prophylaxis for placement of single dental implants. Eur J Oral Implantol. 2009 Winter;2(4):283-92. PMID 20467604
- [Background] Mazzocchi A, Passi L, Moretti R. Retrospective analysis of 736 implants inserted without antibiotic therapy. J Oral Maxillofac Surg. 2007 Nov;65(11):2321-3. doi: 10.1016/j.joms.2007.06.620. PMID 17954332
- [Background] Laskin DM, Dent CD, Morris HF, Ochi S, Olson JW. The influence of preoperative antibiotics on success of endosseous implants at 36 months. Ann Periodontol. 2000 Dec;5(1):166-74. doi: 10.1902/annals.2000.5.1.166. PMID 11885177
- [Background] Choukroun J, Simonpieri A, Del Corso M, Mazor Z, Sammartino G, Dohan Ehrenfest DM. Controlling systematic perioperative anaerobic contamination during sinus-lift procedures by using metronidazole: an innovative approach. Implant Dent. 2008 Sep;17(3):257-70. doi: 10.1097/ID.0b013e318181349a. PMID 18784526
- [Background] Testori T, Drago L, Wallace SS, Capelli M, Galli F, Zuffetti F, Parenti A, Deflorian M, Fumagalli L, Weinstein RL, Maiorana C, Di Stefano D, Valentini P, Gianni AB, Chiapasco M, Vinci R, Pignataro L, Mantovani M, Torretta S, Pipolo C, Felisati G, Padoan G, Castelnuovo P, Mattina R, Del Fabbro M. Prevention and treatment of postoperative infections after sinus elevation surgery: clinical consensus and recommendations. Int J Dent. 2012;2012:365809. doi: 10.1155/2012/365809. Epub 2012 Aug 9. PMID 22927851
- [Background] Esposito M, Cannizzaro G, Bozzoli P, Checchi L, Ferri V, Landriani S, Leone M, Todisco M, Torchio C, Testori T, Galli F, Felice P. Effectiveness of prophylactic antibiotics at placement of dental implants: a pragmatic multicentre placebo-controlled randomised clinical trial. Eur J Oral Implantol. 2010 Summer;3(2):135-43. PMID 20623038
- [Background] Esposito M, Grusovin MG, Loli V, Coulthard P, Worthington HV. Does antibiotic prophylaxis at implant placement decrease early implant failures? A Cochrane systematic review. Eur J Oral Implantol. 2010 Summer;3(2):101-10. PMID 20623035
- [Background] Bratzler DW, Dellinger EP, Olsen KM, Perl TM, Auwaerter PG, Bolon MK, Fish DN, Napolitano LM, Sawyer RG, Slain D, Steinberg JP, Weinstein RA; American Society of Health-System Pharmacists; Infectious Disease Society of America; Surgical Infection Society; Society for Healthcare Epidemiology of America. Clinical practice guidelines for antimicrobial prophylaxis in surgery. Am J Health Syst Pharm. 2013 Feb 1;70(3):195-283. doi: 10.2146/ajhp120568. No abstract available. PMID 23327981
- [Background] Cohen SH, Gerding DN, Johnson S, Kelly CP, Loo VG, McDonald LC, Pepin J, Wilcox MH; Society for Healthcare Epidemiology of America; Infectious Diseases Society of America. Clinical practice guidelines for Clostridium difficile infection in adults: 2010 update by the society for healthcare epidemiology of America (SHEA) and the infectious diseases society of America (IDSA). Infect Control Hosp Epidemiol. 2010 May;31(5):431-55. doi: 10.1086/651706. PMID 20307191
- [Background] Lindeboom JA, van den Akker HP. A prospective placebo-controlled double-blind trial of antibiotic prophylaxis in intraoral bone grafting procedures: a pilot study. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2003 Dec;96(6):669-72. doi: 10.1016/j.tripleo.2003.08.026. PMID 14676756
- [Background] Herzberg R, Dolev E, Schwartz-Arad D. Implant marginal bone loss in maxillary sinus grafts. Int J Oral Maxillofac Implants. 2006 Jan-Feb;21(1):103-10. PMID 16519188
- [Background] Horan TC, Andrus M, Dudeck MA. CDC/NHSN surveillance definition of health care-associated infection and criteria for specific types of infections in the acute care setting. Am J Infect Control. 2008 Jun;36(5):309-32. doi: 10.1016/j.ajic.2008.03.002. No abstract available. PMID 18538699